CLINICAL TRIAL: NCT00478127
Title: Hepatocyte Growth Factor and Cardiovascular Autonomic Function
Status: Completed | Type: Observational
Sponsor: Oita Red Cross Hospital (Other)
Other Study IDs: AO-272
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Last update posted 2007-05-24 (Estimated); Status verified 2007-05

CONDITIONS: Type-2 Diabetes

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
In this study, we tested the hypothesis that elevated HGF is associated with insulin resistance and cardiovascular autonomic dysfunction in type 2 diabetic patients not receiving insulin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type-2 diabetes

Exclusion Criteria:

* Type-1 diabetes

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Futoshi Anan, Principal Investigator — Oita Red Cross Hospital